CLINICAL TRIAL: NCT01094301
Title: A Prospective Multi-Center Pilot Study of the SPR™ System for the Treatment of Post-Stroke Shoulder Pain
Brief Title: Electrical Stimulation for the Treatment of Post-Stroke Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Collaborators: NDI Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NDI-0122-CSP-001
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Shoulder Pain
Keywords: electrical stimulation; neurostimulation; neuromodulation; shoulder pain; post-stroke shoulder pain; hemiplegic shoulder pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- The SPR System (Experimental): The SPR System is an investigational two-staged device which delivers stimulation to the shoulder. Subjects with chronic post-stroke shoulder pain who meet eligibility criteria for the first stage (SPR Trial Stage) will receive a temporary Lead and External Stimulator. Subjects who qualify and who agreed to proceed will advance to the second stage (SPR Implant Stage) which uses an Implantable Pulse Generator (IPG) and Implantable Lead. Subjects will be followed until 36-months after IPG stimulation has been started.
  Interventions: Device: The SPR System

INTERVENTIONS:
Device: The SPR System — The SPR System is an investigational two-staged device which delivers stimulation to the shoulder. Subjects with chronic post-stroke shoulder pain who meet eligibility criteria for the first stage (SPR Trial Stage) will receive a temporary Lead and External Stimulator. Subjects who qualify and who agreed to proceed will advance to the second stage (SPR Implant Stage) which uses an Implantable Pulse Generator (IPG) and Implantable Lead. Subjects will be followed until 36-months after IPG stimulation has been started.

SUMMARY:
Post-stroke shoulder pain is defined as pain in the shoulder area that starts after a person has had a stroke. The SPR System is an investigational device that is being studied for the relief of post-stroke shoulder pain. The SPR System uses electrical stimulation and includes a Trial Stage (where a temporary system is used to see if the subject may benefit from this type of therapy) and may include an Implant Stage (where a small device is implanted under the skin in the chest). The SPR System delivers mild electrical stimulation to the shoulder where the subject feels pain. This research study will evaluate the effect of electrical stimulation on shoulder pain.

Individuals who are over the age of 21, who had a stroke at least six months ago, who experience shoulder pain, and have tried other therapies for their shoulder pain, may be eligible to participate in the first stage of the SPR System. Subjects meeting the specified success criteria at the conclusion of the SPR Trial Stage who experience a return of pain within 6 months of completion of the Trial Stage may be eligible for the second stage (SPR Implant Stage). This research study lasts a little over 3 years and may include 17 visits to the study doctor and at least 8 telephone calls from study staff.

ELIGIBILITY:
Trial Stage Inclusion Criteria:

* At least 21 years of age
* Post-stroke shoulder pain

Trial Stage Exclusion Criteria:

* Use of habit-forming (narcotic) medications
* History of recurrent skin infections
* Bleeding disorder
* Parkinson's Disease, Spinal Cord Injury, traumatic brain injury, Multiple Sclerosis, or complex regional pain syndrome
* Heart arrhythmia or artificial heart valves
* Uncontrolled seizures
* Implanted Electronic Device

Implant Stage Inclusion Criteria

* Had a "return of pain" defined as an increase in pain of at least 2 points compared to the pain intensity score at Visit 5 and has a pain intensity score of at least 4

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Weill Cornell Medical Center, New York, New York
  - Carolinas Healthcare System/Carolinas Rehabilitation, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Moss Rehab/ Albert Einstein Healthcare Network, Elkins Park, Pennsylvania

REFERENCES:
- [Result] Nguyen VQ, Bock WC, Groves CC, Whitney M, Bennett ME, Lechman TE, Strother R, Grill JH, Stager KW, Chae J. Fully implantable peripheral nerve stimulation for the treatment of hemiplegic shoulder pain: a case report. Am J Phys Med Rehabil. 2015 Feb;94(2):146-53. doi: 10.1097/PHM.0000000000000173. PMID 25251248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in April 2010 and was concluded in March 2016. Subjects were screened for the study from the available pool of candidates who presented to the Investigators with shoulder pain following stroke.
Pre-assignment Details: In the original study design, subjects who completed the trial stage and were a success were enrolled in the fully implantable phase. In the revised study design, subjects were required to be both a trial stage success and have a return of pain to be enrolled into the fully implantable phase.
Groups:
- Enrolled Subjects: This group includes subjects that were consented, met eligibility criteria, and received Leads.
Period: Trial Stage
Arm/Group | Enrolled Subjects
Started | 28
Subjects Who Received Smartpatch Lead | 28
Completed | 27
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Implant Stage
Arm/Group | Enrolled Subjects
Started (Trial Stage Subjects who were successful and considered for Implant Stage phase.) | 13
Met Criteria for Implant Stage ((Trial stage success in original design, and a return of pain in the revised design)) | 7
Subjects Who Received SPR IPG | 5
Completed | 5
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — No return of pain | 4

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Type of Stroke [Count of Participants; unit: Participants]
  Hemorrhagic only | 1
  Hemorrhagic and Intracerebral hemorrhage (ICH) | 3
  Intracerebral hemorrhage | 2
  Subarachnoid hemorrhage | 1
  Ischemic only | 20
  Ischemic and Intracerebral hemorrhage (ICH) | 1
Stroke Onset to Enrollment [Mean (Standard Deviation); unit: Years] | 2.7 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity (Trial Stage)
Description: Subjects were asked to report their worst pain score on an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average scores across subjects were reported for Baseline, 3-weeks (End of Placebo), and 6-weeks (End of Treatment).
Time Frame: Baseline, 3-week (Trial Stage), 6-week (Trial Stage)
Population: One subject did not reach end of treatment. Due to this, the subject was not included in the end of treatment analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Trial Stage Subjects: Subjects in the Trial Stage had a Smartpatch Lead placed in the shoulder, used the Smartpatch Peripheral Nerve Stimulation (PNS) System, and received electrical stimulation.
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 28
score on a scale
  Baseline BPI3 Score | 8.2 (1.4)
  End of Placebo BPI3 Score | 6.1 (1.8)
  EOT BPI3 Score: number analyzed (Participants) | 27
  EOT BPI3 Score | 5.0 (2.5)
  Placebo Effect | 2.1 (1.9)
  Treatment Effect: number analyzed (Participants) | 27
  Treatment Effect | 1.0 (2.2)
  Reduction at EOT Compared to Baseline: number analyzed (Participants) | 27
  Reduction at EOT Compared to Baseline | 3.1 (2.4)

2. Primary Outcome: Pain Intensity (Implant Stage)
Description: Subjects were asked to report their worst pain score on an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average scores across subjects were reported for 3-weeks, 6-weeks, 12-weeks, 6-months, 9-months, 12-months, 24-months, and 36 months post IPG-Stim ON.
Time Frame: 3-weeks, 6-weeks, 12-weeks, 6-months, 9-months, 12-months, 24-months, and 36 months post IPG-Stim ON (Implant Stage)
Population: 13 subjects were a trial stage success, 7 of which meet the eligibility criteria for the implant stage, and 5 of the subjects continued on to have the SPR IPG implanted.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant Stage Subjects (Subjects Who Received SPR IPG Implant): Subjects who were a trial stage success in the original study design and who had a return of pain in the revised study design were considered for the Implant Stage. Subjects who were enrolled in this phase had the SPR Implantable Pulse Generator placed in the shoulder and received electrical stimulation.
Arm/Group | Implant Stage Subjects (Subjects Who Received SPR IPG Implant)
Number analyzed (Participants) | 5
score on a scale
  3-weeks post IPG stim-on | 2.0 (1.3)
  6-weeks post IPG stim-on | 0.3 (0.8)
  12-weeks post IPG stim-on | 0.4 (0.9)
  6-months post IPG stim-on | 1.6 (1.8)
  9-months post IPG stim-on | 0.6 (1.3)
  12-months post IPG stim-on | 0.8 (1.3)
  24-months post IPG stim-on | 1.6 (3.0)
  36-months post IPG stim-on | 1.2 (1.6)

3. Primary Outcome: Device-Related Adverse Events
Description: At each study visit following the baseline assessment at Visit 1, subjects were questioned if any changes in their medical status or condition had occurred since their previous visit. If the subject experienced a change that was an adverse event, an Adverse Event Form was completed by the site. The number of subjects that experienced at least one study-related adverse event is reported here.
Time Frame: Total of 86 months (from when the first subjects enrolled to when the last subject completed the study)
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 28
Participants
  Subjects who reported device related AEs | 20
  Subjects who did not report any device related AEs | 8

4. Primary Outcome: Number of Subjects Who Were a Trial Stage Success
Description: The number of subjects who were a trial stage success is presented. Trial Stage Success for each subject was determined by a 2-point reduction in Brief Pain Inventory question 3 at the end of t.he Trial Stage beyond any placebo effect.
Time Frame: End of Treatment (EOT)
Population: Twenty-seven subjects completed the study through end of treatment (EOT)
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 27
Participants | 13

5. Primary Outcome: Number of Subjects Who Were an Implant Stage Success
Description: Number of subjects who were an Implant Stage Success is presented. Implant Stage Success for each subject was determined by a 2-point reduction in Brief Pain Inventory question 3 at 12-week post IPG stimulation ON beyond any placebo effect.
Time Frame: 12-weeks post IPG-Stim ON
Measure: Count of Participants; unit: Participants
Arm/Group | Implant Stage Subjects (Subjects Who Received SPR IPG Implant)
Number analyzed (Participants) | 5
Participants | 5

6. Secondary Outcome: Pain Interference (Trial Stage)
Description: Subjects were asked to rate the degree to which their pain has interfered with general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life on an 11-point numerical rating scale where 0 represents "does not interfere" and 10 represents "completely interferes." The average scores across subjects were reported for Baseline, 3-weeks (End of Placebo), and 6-weeks (End of Treatment).
Time Frame: Baseline, 3-week (Trial Stage), 6-week (Trial Stage)
Population: One subject did not reach end of treatment and was not included in the end of treatment analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 28
score on a scale
  Baseline BPI9 Score | 6.2 (2.5)
  End of Placebo BPI9 Score | 4.7 (2.3)
  EOT BPI9 Score: number analyzed (Participants) | 27
  EOT BPI9 Score | 3.2 (3.0)
  BPI9 Reduction at EOT Compared to End of Placebo: number analyzed (Participants) | 27
  BPI9 Reduction at EOT Compared to End of Placebo | 1.3 (2.1)
  BPI9 Reduction at EOT Compared to Baseline: number analyzed (Participants) | 27
  BPI9 Reduction at EOT Compared to Baseline | 2.9 (2.9)

7. Secondary Outcome: Pain-Free Passive Range of Motion (Trial Stage)
Description: Pain-Free Passive Range of Motion (ROM) was assessed. The average ROMs for all subjects were reported for Baseline, 3-weeks (End of Placebo), and 6-weeks (End of Treatment).
Time Frame: Baseline, 3-week (Trial Stage), 6-week (Trial Stage);
Population: One subject did not reach end of treatment and was not included in the end of treatment analysis.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 28
Degrees
  Baseline ROM | 89.8 (53.1)
  End of Placebo ROM | 102.8 (49.0)
  EOT ROM: number analyzed (Participants) | 27
  EOT ROM | 119.5 (38.6)
  Increase in ROM at EOT Compared to End of Placebo: number analyzed (Participants) | 27
  Increase in ROM at EOT Compared to End of Placebo | 17.5 (41.3)
  Increase in ROM at EOT Compared to Baseline: number analyzed (Participants) | 27
  Increase in ROM at EOT Compared to Baseline | 31.2 (51.7)

8. Secondary Outcome: Quality of Life (Trial Stage)
Description: Subjects were asked to complete the Short Form Health Survey Version 2 (SF-36v2) to assess basic physical functioning and emotional well-being regardless of the disease or treatment. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. The eight domains are physical functioning, role limitations due to physical problems, social functioning, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perceptions. The mean scores for Baseline, 3-week (End of Placebo), and 6-week (End of Treatment) were reported.
Time Frame: Baseline, 3-week (Trial Stage), 6-week (Trial Stage)
Population: Computer analysis of the available data was not completed for four subjects at baseline, six subjects at 3-weeks, and eight subjects at end of treatment. Additionally, one subject did not reach end of treatment and was not included in the end of treatment analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 24
Scores on a scale
  Bodily Pain; Baseline | 32.2 (5.7)
  Bodily Pain; 3-week (Trial Stage): number analyzed (Participants) | 22
  Bodily Pain; 3-week (Trial Stage) | 36.2 (6.3)
  Bodily Pain; 6-week (Trial Stage): number analyzed (Participants) | 19
  Bodily Pain; 6-week (Trial Stage) | 39.4 (7.0)
  Bodily Pain; Change from End of Sham to EOT: number analyzed (Participants) | 19
  Bodily Pain; Change from End of Sham to EOT | 3.4 (5.7)
  Role-physical; Baseline | 29.8 (8.4)
  Role-physical; 3-week (Trial Stage): number analyzed (Participants) | 22
  Role-physical; 3-week (Trial Stage) | 30.7 (10.3)
  Role-physical; 6-week (Trial Stage): number analyzed (Participants) | 19
  Role-physical; 6-week (Trial Stage) | 33.6 (9.1)
  Role-physical; Change from End of Sham to EOT: number analyzed (Participants) | 19
  Role-physical; Change from End of Sham to EOT | 2.9 (5.6)
  Role-emotional; Baseline | 35.7 (14.6)
  Role-emotional; 3-week (Trial Stage): number analyzed (Participants) | 22
  Role-emotional; 3-week (Trial Stage) | 34.2 (15.7)
  Role-emotional; 6-week (Trial Stage): number analyzed (Participants) | 19
  Role-emotional; 6-week (Trial Stage) | 38.6 (13.6)
  Role-emotional; Change from End of Sham to EOT: number analyzed (Participants) | 19
  Role-emotional; Change from End of Sham to EOT | 3.0 (9.8)
  Mental health; Baseline | 43.1 (11.5)
  Mental health; 3-week (Trial Stage): number analyzed (Participants) | 22
  Mental health; 3-week (Trial Stage) | 44.8 (11.7)
  Mental health; 6-week (Trial Stage): number analyzed (Participants) | 19
  Mental health; 6-week (Trial Stage) | 48.5 (9.4)
  Mental health; Change from End of Sham to EOT: number analyzed (Participants) | 19
  Mental health; Change from End of Sham to EOT | 3.5 (7.6)
  Physical functioning; Baseline | 27.3 (9.6)
  Physical functioning; 3-week (Trial): number analyzed (Participants) | 22
  Physical functioning; 3-week (Trial) | 27.3 (11.2)
  Physical functioning; 6-week (Trial Stage): number analyzed (Participants) | 19
  Physical functioning; 6-week (Trial Stage) | 29.6 (11.2)
  Physical functioning; Change from EOS to EOT: number analyzed (Participants) | 19
  Physical functioning; Change from EOS to EOT | 2.5 (5.3)
  Social functioning; Baseline | 39.6 (12.5)
  Social functioning; 3-week (Trial Stage): number analyzed (Participants) | 22
  Social functioning; 3-week (Trial Stage) | 39.3 (12.9)
  Social functioning; 6-week (Trial Stage): number analyzed (Participants) | 19
  Social functioning; 6-week (Trial Stage) | 43.9 (10.2)
  Social functioning; Change from End of Sham to EOT: number analyzed (Participants) | 19
  Social functioning; Change from End of Sham to EOT | 3.1 (8.8)
  Vitality; Baseline | 45.5 (7.2)
  Vitality; 3-week (Trial Stage): number analyzed (Participants) | 22
  Vitality; 3-week (Trial Stage) | 45.4 (8.0)
  Vitality; 6-week (Trial Stage): number analyzed (Participants) | 19
  Vitality; 6-week (Trial Stage) | 48.0 (8.6)
  Vitality; Change from End of Sham to EOT: number analyzed (Participants) | 19
  Vitality; Change from End of Sham to EOT | 1.9 (6.6)
  General Health; Baseline | 42.4 (11.0)
  General Health; 3-week (Trial Stage): number analyzed (Participants) | 22
  General Health; 3-week (Trial Stage) | 39.9 (8.6)
  General Health; 6-week (Trial Stage): number analyzed (Participants) | 19
  General Health; 6-week (Trial Stage) | 41.1 (9.0)
  General Health; Change from End of Sham to EOT: number analyzed (Participants) | 19
  General Health; Change from End of Sham to EOT | 1.0 (6.6)

9. Secondary Outcome: Number of Participants Completing the Economic Impact Survey
Description: Subjects were asked to document pain medication, doctor visits, supplies, related treatments, need for caregivers, time spent in skilled nursing facilities, and lost work due to their shoulder pain. This data was collected from subjects at Baseline and asked to recall this data for the 6-months prior to study enrollment. National average costs were not available for these data points, and therefore the overall economic impact of shoulder pain could not be reported.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 28
Participants
  Subjects who completed economic impact survey | 25
  Subjects not completing economic impact survey | 3

10. Secondary Outcome: Emotional Functioning (Trial Stage)
Description: Subjects were asked to complete the Beck Depression Inventory Version 2 (BDI-II), a 21 question survey to assess depressive symptoms. Each answer was scored on a scale value of 0 to 3 and a sum was taken for all 21 questions. Higher total scores indicated more severe depressive symptoms. The standardized cutoffs used were: 0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, and 29-63: severe depression. Mean BDI-II scores were calculated across subjects and were reported for Baseline, 3-weeks (End of Placebo), and 6-weeks (End of Treatment).
Time Frame: Baseline, 3-week (Trial Stage), 6-week (Trial Stage)
Population: One subject did not reach end of treatment and was not included in the end of treatment analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 28
Scores on a scale
  Baseline BDI-II Score | 13.4 (8.8)
  End of Placebo BDI-II Score | 14.8 (10.0)
  EOT BDI-II Score: number analyzed (Participants) | 27
  EOT BDI-II Score | 12.9 (9.9)
  BDI-II Reduction at EOT Compared to End of Placebo: number analyzed (Participants) | 27
  BDI-II Reduction at EOT Compared to End of Placebo | 1.6 (6.9)
  BDI-II Reduction at EOT Compared to Baseline: number analyzed (Participants) | 27
  BDI-II Reduction at EOT Compared to Baseline | 0 (7.1)

11. Secondary Outcome: User Satisfaction (Trial Stage)
Description: Subjects completed a sponsor-developed survey with questions pertaining to their feelings about the Smartpatch Stimulation System as a method for managing post-stroke shoulder pain.
Time Frame: 6-week (Trial Stage)
Population: This survey was not a part of the original study design. It was administered to 21 subjects. Additionally, one subject did not answer the questions related to their study experience.
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 20
Participants
  Reported study had positive impact on their life | 18
  Reported being satisfied with experience in study | 19
  Would recommend participation in study to a friend | 20

12. Secondary Outcome: Global Impact of Stimulation Therapy (Trial Stage)
Description: The Patient Global Impression of Change asks subjects to rate their improvement with treatment on a 7-point scale ranging from "very much worse" to "very much improved". The subjects combine all the components of their experience into one overall score.
Time Frame: 3-week (Trial Stage), 6-week (Trial Stage)
Population: One subject did not reach end of treatment and was not included in the 6-week treatment analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 28
Participants
  3-week (Trial Stage): Very much worse | 0
  3-week (Trial Stage): Much worse | 0
  3-week (Trial Stage): Minimally worse | 0
  3-week (Trial Stage): No Change | 5
  3-week (Trial Stage): Minimally improved | 17
  3-week (Trial Stage): Much improved | 4
  3-week (Trial Stage): Very much improved | 2
  6-week (Trial Stage): number analyzed (Participants) | 27
  6-week (Trial Stage): Very much worse | 0
  6-week (Trial Stage): Much worse | 0
  6-week (Trial Stage): Minimally worse | 0
  6-week (Trial Stage): No Change | 3
  6-week (Trial Stage): Minimally improved | 10
  6-week (Trial Stage): Much improved | 13
  6-week (Trial Stage): Very much improved | 1

13. Secondary Outcome: Quality of Life (Implant Stage)
Description: Subjects were asked to complete the Short Form Health Survey Version 2 (SF-36v2) to assess basic physical functioning and emotional well-being regardless of the disease or treatment. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. The eight domains are physical functioning, role limitations due to physical problems, social functioning, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perceptions. The mean scores for 3-weeks, 12-weeks, 6-months, 9-months, and 12-months, post IPG-Stim ON were reported.
Time Frame: 3-weeks, 12-weeks, 6-months, 9-months, 12-months post IPG-Stim ON (Implant Stage)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Implant Stage Subjects (Subjects Who Received SPR IPG Implant)
Number analyzed (Participants) | 5
Scores on a scale
  Bodily pain; 3-weeks (Implant) | 42.6 (5.0)
  Bodily pain; 12-weeks (Implant Stage) | 46.7 (10.5)
  Bodily pain; 6-months (Implant Stage) | 45.1 (4.6)
  Bodily pain; 9-months (Implant Stage) | 43.7 (11.5)
  Bodily pain; 12-months (Implant Stage) | 50.1 (7.8)
  Role-physical; 3-weeks (Implant Stage) | 38.3 (9.5)
  Role-physical; 12-weeks (Implant Stage) | 35.1 (10.7)
  Role-physical; 6-months (Implant Stage | 40.4 (6.6)
  Role-physical; 9-months (Implant Stage | 37.1 (14.4)
  Role-physical; 12-months (Implant Stage | 37.5 (10.0)
  Role-emotional; 3-weeks (Implant Stage) | 47.4 (7.8)
  Role-emotional; 12-weeks (Implant Stage) | 38.3 (15.7)
  Role-emotional; 6-months (Implant Stage) | 47.4 (13.2)
  Role-emotional; 9-months (Implant Stage) | 39.8 (13.2)
  Role-emotional; 12-months (Implant Stage) | 43.6 (15.5)
  Mental health; 3-weeks (Implant Stage) | 52.4 (5.2)
  Mental health; 12-weeks (Implant Stage) | 49.0 (7.7)
  Mental health; 6-months (Implant Stage) | 50.7 (9.1)
  Mental health; 9-months (Implant Stage) | 46.8 (10.9)
  Mental health; 12-months (Implant Stage) | 47.9 (12.8)
  Physical functioning; 3-weeks (Implant Stage) | 32.1 (15.1)
  Physical functioning; 12-weeks (Implant Stage) | 31.3 (13.0)
  Physical functioning; 6-months (Implant Stage) | 31.3 (13.2)
  Physical functioning; 9-months (Implant Stage) | 32.1 (13.8)
  Physical functioning; 12-months (Implant Stage) | 24.8 (19.5)
  Social functioning; 3-weeks (Implant Stage) | 43.5 (2.9)
  Social functioning; 12-weeks (Implant Stage) | 46.7 (5.9)
  Social functioning; 6-months (Implant Stage) | 47.8 (8.2)
  Social functioning; 9-months (Implant Stage) | 45.6 (10.8)
  Social functioning; 12-months (Implant Stage) | 44.6 (12.3)
  Vitality; 3-weeks (Implant Stage) | 48.4 (2.5)
  Vitality; 12-weeks (Implant Stage) | 49.6 (5.4)
  Vitality; 6-months (Implant Stage) | 51.4 (5.4)
  Vitality; 9-months (Implant Stage) | 49.6 (13.3)
  Vitality; 12-months (Implant Stage) | 50.2 (9.6)
  General health; 3-weeks (Implant Stage) | 39.7 (7.2)
  General health; 12-weeks (Implant Stage) | 40.1 (8.0)
  General health; 6-months (Implant Stage) | 41.7 (8.2)
  General health; 9-months (Implant Stage) | 41.3 (11.6)
  General health; 12-months (Implant Stage) | 38.0 (15.3)

14. Secondary Outcome: Pain Interference (Implant Stage)
Description: Subjects were asked to rate the degree to which their pain has interfered with general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life on an 11-point numerical rating scale where 0 represents "does not interfere" and 10 represents "completely interferes." The average scores across subjects were reported for 3-weeks, 6-weeks, 12-weeks, 6-months, 9-months, and 12-months post IPG-Stim On.
Time Frame: 3-weeks, 6-weeks, 12-weeks, 6-months, 9-months, 12-months post IPG-Stim ON (Implant Stage)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implant Stage Subjects (Subjects Who Received SPR IPG Implant)
Number analyzed (Participants) | 5
score on a scale
  3-weeks post IPG stim-on | 0.5 (0.4)
  6-weeks post IPG stim-on | 0.1 (0.2)
  12-weeks post IPG stim-on | 0.2 (0.4)
  6-months post IPG stim-on | 0.3 (0.5)
  9-months post IPG stim-on | 0.1 (0.2)
  12-months post IPG stim-on | 0.1 (0.3)
  24-months post IPG stim-on | 0.4 (0.8)
  36-months post IPG stim-on | 0.0 (0.1)

15. Secondary Outcome: Pain-Free Passive Range of Motion (Implant Stage)
Description: Pain-Free Passive Range of Motion (ROM) was assessed. The average ROMs for all subjects were reported for 3-weeks, 12-weeks, 6-months, 9-months, and 12-months post IPG-Stim ON.
Time Frame: 3-weeks, 12-weeks, 6-months, 9-months, 12-months post IPG-Stim ON (Implant Stage)
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Implant Stage Subjects (Subjects Who Received SPR IPG Implant)
Number analyzed (Participants) | 5
Degrees
  3-weeks post IPG stim-on | 125.2 (25.7)
  12-weeks post IPG stim-on | 119.8 (11.6)
  6-months post IPG stim-on | 141.2 (17.5)
  9-months post IPG stim-on | 146.6 (20.3)
  12-months post IPG stim-on | 151.4 (14.6)

16. Secondary Outcome: Emotional Functioning (Implant Stage)
Description: Subjects were asked to complete the Beck Depression Inventory Version 2 (BDI-II), a 21 question survey to assess depressive symptoms. Each answer was scored on a scale value of 0 to 3 and a sum was taken for all 21 questions. Higher total scores indicated more severe depressive symptoms. The standardized cutoffs used were: 0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, and 29-63: severe depression. Mean BDI-II scores were calculated across subjects and were reported for 3-weeks, 12-weeks, 6-months, 9-months, and 12-months post IPG-Stim ON.
Time Frame: 3-weeks, 12-weeks, 6-months, 9-months, 12-months post IPG-Stim ON (Implant Stage)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Implant Stage Subjects (Subjects Who Received SPR IPG Implant)
Number analyzed (Participants) | 5
Scores on a scale
  3-weeks post IPG stim-on | 10.2 (9.7)
  12-weeks post IPG stim-on | 8.4 (7.7)
  6-months post IPG stim-on | 10.6 (10.1)
  9-months post IPG stim-on | 12.4 (12.6)
  12-months post IPG stim-on | 12.6 (15)

17. Secondary Outcome: Global Impact of Stimulation Therapy (Implant Stage)
Description: as for outcome 12
Time Frame: 3-weeks, 12-weeks, 6-months, 9-months, 12-months, 24-months, and 36-months Post IPG-Stim ON (Implant Stage)
Measure: Count of Participants; unit: Participants
Arm/Group | Implant Stage Subjects (Subjects Who Received SPR IPG Implant)
Number analyzed (Participants) | 5
Participants
  3-weeks (Implant Stage): Very much worse | 0
  3-weeks (Implant Stage): Much worse | 0
  3-weeks (Implant Stage): Minimally worse | 0
  3-weeks (Implant Stage): No change | 0
  3-weeks (Implant Stage): Minimally improved | 3
  3-weeks (Implant Stage): Much improved | 1
  3-weeks (Implant Stage): Very much improved | 1
  12-weeks (Implant Stage): Very much worse | 0
  12-weeks (Implant Stage): Much worse | 0
  12-weeks (Implant Stage): Minimally worse | 0
  12-weeks (Implant Stage): No change | 0
  12-weeks (Implant Stage): Minimally improved | 1
  12-weeks (Implant Stage): Much improved | 3
  12-weeks (Implant Stage): Very much improved | 1
  6-months (Implant Stage): Very much worse | 0
  6-months (Implant Stage): Much worse | 0
  6-months (Implant Stage): Minimally worse | 0
  6-months (Implant Stage): No change | 0
  6-months (Implant Stage): Minimally improved | 0
  6-months (Implant Stage): Much improved | 4
  6-months (Implant Stage): Very much improved | 1
  9-months (Implant Stage): Very much worse | 0
  9-months (Implant Stage): Much worse | 0
  9-months (Implant Stage): Minimally worse | 0
  9-months (Implant Stage): No change | 0
  9-months (Implant Stage): Minimally improved | 0
  9-months (Implant Stage): Much improved | 4
  9-months (Implant Stage): Very much improved | 1
  12-months (Implant Stage): Very much worse | 0
  12-months (Implant Stage): Much worse | 0
  12-months (Implant Stage): Minimally worse | 0
  12-months (Implant Stage): No change | 0
  12-months (Implant Stage): Minimally improved | 1
  12-months (Implant Stage): Much improved | 3
  12-months (Implant Stage): Very much improved | 1
  24-months (Implant Stage): Very much worse | 0
  24-months (Implant Stage): Much worse | 0
  24-months (Implant Stage): Minimally worse | 0
  24-months (Implant Stage): No change | 0
  24-months (Implant Stage): Minimally improved | 0
  24-months (Implant Stage): Much improved | 3
  24-months (Implant Stage): Very much improved | 2
  36-months (Implant Stage): Very much worse | 0
  36-months (Implant Stage): Much worse | 0
  36-months (Implant Stage): Minimally worse | 0
  36-months (Implant Stage): No change | 1
  36-months (Implant Stage): Minimally improved | 0
  36-months (Implant Stage): Much improved | 2
  36-months (Implant Stage): Very much improved | 2

18. Secondary Outcome: User Satisfaction (Implant Stage)
Description: Subjects completed a sponsor-developed survey with questions pertaining to their feelings about the IPG System as a method for managing post-stroke shoulder pain.
Time Frame: 12-weeks,12-months post IPG-Stim ON (Implant Stage)
Measure: Count of Participants; unit: Participants
Arm/Group | Implant Stage Subjects (Subjects Who Received SPR IPG Implant)
Number analyzed (Participants) | 5
Participants
  Satisfied with experience 12-weeks Implant Stage | 5
  Satisfied with experience 12-mths Implant Stage | 5
  Pleased with the SPR System 12-wks Implant Stage | 5
  Pleased with the SPR System 12-mths Implant Stage | 5
  Would recommend to a friend 12-wks Implant Stage | 5
  Would recommend to a friend 12-mths Implant Stage | 5
  Wanted to participate again 12-wks Implant Stage | 5
  Wanted to participate again 12-mnths Implant Stage | 5
  Positive impact on life 12-wks Implant Stage | 5
  Positive impact on life 12-mnths Implant Stage | 5

19. Secondary Outcome: Reduction in Arm Impairment and Improvement in Activities of Daily Living (Trial Stage)
Description: Subjects were asked to assess their arm impairment using the Stroke Upper Limb Capacity Scale (SULCS) test. The SULCS is a validated upper limb capacity scale which includes tasks directly related to activities of daily living individuals experience in their home environment. The SULCS consists of 10 items, with each item having a possible score of 0 or 1: 3 items for arm capacity without active hand capacity; 4 items for arm capacity and basic hand capacity; and, 3 items for complex hand capacity. These scores were summed with a higher score indicating better capacity, with 10 being the max score. The average score across subjects were reported for Baseline, 3-weeks (End of Placebo), and 6-weeks (End of Trial Stage).
Time Frame: Baseline, 3-week (Trial Stage), 6-week (Trial Stage)
Population: This survey was collected for the last 9 subjects enrolled in the Trial Stage due to a mid-study protocol change. Of these 9 subjects,6 subjects completed the survey at 3-weeks and 8 subjects completed the survey at 6-weeks.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Trial Stage Subjects
Number analyzed (Participants) | 9
Scores on a scale
  Baseline SULCS Score | 3.8 (3.7)
  3-weeks SULCS Score (Trial Stage): number analyzed (Participants) | 6
  3-weeks SULCS Score (Trial Stage) | 3.7 (3.4)
  6-weeks SULCS Score (Trial Stage): number analyzed (Participants) | 8
  6-weeks SULCS Score (Trial Stage) | 3.3 (3.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 86 months (time from when the first subject was enrolled in 5/27/10 to when the last subject was completed in 7/25/17).
Description: At each study visit following the baseline assessment, subjects were questioned if any changes in their medical status or condition had occurred. If the change was an adverse event, an adverse event form was completed by the site.
Arm/Group | Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 24/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=28)
Complaints of Chest Pain (Cardiac disorders) | 1 (2) — One event was not study-related, and the relationship of one was unable to be determined
Myocardial Infarction (Cardiac disorders) | 1 (1) — Not study-related
Acute heart failure exacerbation (Cardiac disorders) | 1 (1) — Not study-related
Syncope (Cardiac disorders) | 3 (4) — Not study-related
Cellulitis (Infections and infestations) | 1 (1) — Not study-related
Seizure (Nervous system disorders) | 2 (2) — Not study-related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=28)
Skin Irritation (redness, mild skin abrasion, or mild grade 1 pressure sore with intact skin) (Skin and subcutaneous tissue disorders) | 11 (12) — Eleven were Study-related, and one was unrelated
Painful Stimulation (Product Issues) | 4 (7) — Six were study-related, and the relationship of one was unable to be determined
Painful Keloid (Skin and subcutaneous tissue disorders) | 1 (1) — Study-related
Granuloma (Skin and subcutaneous tissue disorders) | 5 (5) — Study-related
Distress (Psychiatric disorders) | 1 (1) — Study-related
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) — Study-related
Tenderness at lead exit site (Skin and subcutaneous tissue disorders) | 1 (1) — Study-related
Fall (General disorders) | 4 (5) — Not study-related
Migraines (Nervous system disorders) | 1 (1) — Not study-related
Nerve Pain (Nervous system disorders) | 1 (1) — Not study-related
Atypical sensation (Tingling/Quivering of fingers/hands or "shock-like" episode after lead removal) (General disorders) | 3 (3) — One was not study-related and the other two were unable to be determined
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not study-related
Subconjunctival hematoma (General disorders) | 1 (1) — Not study-related
Vomiting (General disorders) | 1 (1) — Not study-related
Malaise (General disorders) | 1 (1) — Not study-related
Total body aches (General disorders) | 1 (1) — Not study-related
Ipsilateral spasms of upper arm and shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — Not study-related
Report of redness on hand (Skin and subcutaneous tissue disorders) | 1 (1) — Not study-related
Elbow stiffness and appearance of fluid (Musculoskeletal and connective tissue disorders) | 1 (1) — Not study-related
Benign tumor index finger (Skin and subcutaneous tissue disorders) | 1 (1) — Not study-related
Release of achilles tendon (Surgical and medical procedures) | 1 (1) — Not study-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT01094301/Prot_SAP_000.pdf